CLINICAL TRIAL: NCT06557395
Title: UNMET NURSING CARE PERCEPTIONS OF INTENSIVE CARE NURSES: A QUALITATIVE STUDY
Brief Title: UNMET CARE PERCEPTIONS OF INTENSIVE CARE NURSES
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Dilek KIYMAZ, Lecturer Dr., Ondokuz Mayıs University
Other Study IDs: UNMET NURSING CARE PERCEPTIONS
Record Dates: First submitted 2024-08-07; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Nurse's Role
Keywords: care perception, patient, nurse, unmet care, intensive care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted to determine the perceptions of intensive care nurses regarding unmet care. A qualitative descriptive approach. The study was completed between April and September 2023 by conducting semi-structured individual interviews with 20 intensive care nurses in a Training and Research Hospital in Turkey and analyzed using the inductive content analysis method.

DETAILED DESCRIPTION:
Unmet nursing care may occur due to systemic, institutional or nursing-related reasons. Reasons such as insufficient staff and equipment, excessive workload (Pereira et al., 2020), confusion between disciplines, and failure to prioritize care play an important role in missed care (Chaboyer et al., 2021; Dutra & Guirardello, 2021; Kılıç et al., 2023). In summary, while improvements should be made in nursing care practices to ensure patient safety and quality of care, systemic improvements should also be made. In order to make these improvements, it should be determined what the missed nursing care experienced and perceived in the clinical field is and what causes them. This research was conducted to determine the perceptions of intensive care nurses about unmet nursing care. This study is a qualitative design research conducted with intensive care nurses. In the study, a purposeful sample selection was made in accordance with the qualitative research approach. The number of participants was determined according to data saturation and is based on the volunteering of a total of 20 intensive care nurses. During the interview, the participants were asked a personal information form and expert opinion on the subject, as well as in-depth interview questions in a semi-structured information form consisting of eight questions.

ELIGIBILITY:
Inclusion Criteria:

* working in intensive care
* volunteering to participate in the study

Exclusion Criteria:

* not volunteering to participate in the study

Ages: 23 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study comprised research with qualitative design completed with intensive care nurses.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
What is the perception of care among intensive care nurses? | April-September 2023
  This study is a qualitative design study conducted with intensive care nurses. In the study, a purposeful sampling method was used in accordance with the qualitative research approach. The number of participants was determined according to data saturation and was based on the voluntary participation of a total of 20 intensive care nurses. During the interview, participants were asked to fill out a personal information form and expert opinions on the subject, as well as in-depth interview questions in a semi-structured information form consisting of eight questions. Data were collected through face-to-face individual interviews with nurses working in the intensive care unit of a Training and Research Hospital between April and September 2023. In-depth interview questions were prepared in line with literature knowledge and expert opinions were obtained.
What are the thoughts of intensive care nurses regarding the perception of unmet care? | April-September 2023
  After the interviews were completed, the raw data were manually transcribed by the researchers. The content analysis method was used in the evaluation of the data. The data were read several times by the researchers and codes were created from each word, sentence and paragraph. The analysis of the data was carried out manually using the level coding system and themes were created. Level coding was applied as open coding (first level), selective coding (second level), themes (third level) (Yıldırım & Şimşek 2016). After this stage, the relevant codes were classified and themes and sub-themes were created (Elo & Kyngäs, 2008; Vaismoradi et al., 2013).

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No